CLINICAL TRIAL: NCT04988282
Title: Systemic Corticosteroids in Treatment of Post-COVID-19 Interstitial Lung Disease
Acronym: STERCOV-ILD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Turkish Thoracic Society (Other)
Responsible Party: Principal Investigator, Metin Akgun, MD, Professor, Turkish Thoracic Society
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STERCOV-ILD
Record Dates: First submitted 2021-07-22; First posted 2021-08-03 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Covid19; COVID-19 Pneumonia; Interstitial Lung Disease
MeSH Terms: conditions — COVID-19; Lung Diseases, Interstitial | interventions — Methylprednisolone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Steroid (Active Comparator): Methylprednisolone, oral, 0.5 mg/kg/day, 4 weeks; followed by a gradual reduction of 25% every 2 weeks.
  Total Duration:12-16 weeks
  Interventions: Drug: Methylprednisolone Tablet
- control (Other): standard symptom-relief therapy (since there is no current standard therapy for post-COVID Interstitial Lung Disease, patients in this arm will be commenced symptom-relief therapies including bronchodilators, inhaled corticosteroids, non-steroid anti-inflammatories, cough relievers, and long-term oxygen if the patient has respiratory failure)
  Interventions: Drug: Methylprednisolone Tablet

INTERVENTIONS:
Drug: Methylprednisolone Tablet — Methylprednisolone, oral, 0.5 mg/kg/day, 4 weeks
  Other Names: Prednol

SUMMARY:
Aim: To investigate the efficacy of systemic corticosteroids in treatment for Post-COVID-19 Interstitial Lung Disease.

Method: Method: In this multi-centre, prospective, randomised controlled open label clinical trial, patients are divided into two arms: standard treatment arm and standard plus systemic corticosteroid arm. After twelve weeks; clinical, functional, and radiological improvement will being assessed as primary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Post-COVID-19 Interstitial Lung Disease (ILD) patients who had completed the treatment of acute phase and have recovered, but despite after 90 days from recovery diagnosed as post-COVID ILD based upon the persistent respiratory symptoms with functional impairment and radiological sequela.

  * At least 90 days required after discharge for hospitalized patients or termination of isolation for outpatients
* Confirmation of the diagnosis of COVID-19 via real time polymerase chain reaction assay (rt-PCR) or antigen or antibody test in the acute phase of COVID-19.
* Presence of sequelae interstitial changes in follow-up (pre-enrollment) thorax high-resolution computed tomography (HRCT)/CT.
* Presence of persistent respiratory symptoms in the post-COVID-19 period or hypoxemia at rest and/or desaturation with exercise.

Exclusion Criteria:

* Patients who had a normal lung imaging examination (radiography, tomography, etc.) at discharge or enrollment phase
* Pre-existing diffuse parenchymal lung disease before pandemic
* Cystic bronchiectasis
* Presence of contraindications for systemic corticosteroids (uncontrolled Diabetes, uncontrolled Hypertension, unstable angina pectoris, history of acute coronary syndrome at last month, presence of active infection, active peptic ulcer, presence of uncontrolled psychiatric disease, etc.)
* Decompensated heart failure
* Contraindications for pulmonary function tests and those who cannot cooperate with the test
* Younger than 18 years old
* Pregnant women
* Breastfeeding women
* Those who do not give written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
% of patients with clinical improvement | 12 weeks
  Clinical improvement is identified as grade 0 modified Medical Research Council (mMRC) dyspnea score with no respiratory complaints.
% of patients with functional improvement | 12 weeks
  A combination of following features: Sp02 is greater than 95% at rest; No desaturation during 6MWT; FVC is greater than 80%; DLCO is greater than 80%
% of patients with radiological improvement | 12 weeks
  At least 50% regression in extension of interstitial lesions on thorax CT. (Thorax CT images will be assessed by a radiologist and a pulmonologist who is expertised in thoracic CT.)

SECONDARY OUTCOMES:
Improvement of diffusion capacity of lung for carbon monoxide (DLCO) | 12 weeks
  Percentage of increase in diffusion capacity of lung for carbon monoxide
Improvement of Forced Vital Capacity (FVC) | 12 weeks
  Change in Forced Vital Capacity
Improvement of arterial oxygen saturation (SaO2) | 12 weeks
  Change in Oxygen Saturation at room air
Improvement of Exercise Capacity | 12 weeks
  Change in 6 minute walking test duration
Improvement of mMRC dyspnea score | 12 weeks
  Change in mMRC dyspnea score
Respiratory-cause emergency visit and hospitalisation | 12 weeks
  Number of patients who had respiratory-cause emergency visit and hospitalization during study period.
Mortality rate | 12 weeks
  Mortality rate
Advers events | 12 weeks
  Systemic corticosteroid related advers events

CONTACTS AND LOCATIONS:
Overall Officials: METİN AKGÜN, Study Director — ATATURK UNIVERSITY FACULTY OF MEDICINE
Locations (1):
- Ufuk University Medicine Faculty, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No